CLINICAL TRIAL: NCT05450913
Title: Frequency of Piriformis Syndrome in Hip and/or Leg Pain: Does the Presence of One Pathology Rule Out the Other?
Brief Title: Frequency of Piriformis Syndrome:Does the Presence of One Pathology Rule Out the Other?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, MD, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: piriformis
Record Dates: First submitted 2022-03-21; First posted 2022-07-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
Keywords: piriformis syndrome; myofascial pain; ultrasound guidance; trigger point injection
MeSH Terms: conditions — Chronic Pain; Piriformis Muscle Syndrome | interventions — Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with unilateral hip and leg pain (Other): Musculoskeletal system examination, neurological examination, visual analog scale (VAS) score and DN4 (Douleur Neuropathique 4 Questions) of patients presenting with unilateral hip and/or leg pain, 3 tests frequently used in the diagnosis of priformis (Freiberg test, Pace sign, FADIR) ) will be applied.
  Patients with suspected priformis syndrome will be given an intramuscular injection If the pain intensity decreases by 50% or more after the intramuscular injection, the diagnosis of piriformis will be made.
  Interventions: Drug: Priformis intramuscular injection with %2 lidocain

INTERVENTIONS:
Drug: Priformis intramuscular injection with %2 lidocain — Priformis intramuscular injection will be administered with 5 cc 2% lidocaine, accompanied by a nerve stimulator under ultrasound guidance
  Other Names: pyriformis intramuscular injection or diagnostic test with local anesthetic

SUMMARY:
The purpose of the investigators is to determine the frequency of priformis syndrome in patients presenting with hip and/or leg pain and to investigate the association of Priformis syndrome with other pathologies of the lumbar spine and hip.

DETAILED DESCRIPTION:
Priformis Syndrome is a neuromuscular disorder characterized by compression or irritation of the sciatic nerve under the piriformis muscle, tenderness in the piriformis muscle, and back, hip, and leg pain. The pain may radiate along the sciatic nerve trace in the gluteal region and posterior thigh. Diagnosis is based on clinical symptoms, specific physical examination findings, and positive response to local injection.

The diagnosis of piriformis syndrome is usually made only after lumbar spine pathologies are excluded. This traditional approach leads to underdiagnosis of piriformis syndrome. More than one cause may coexist in hip and/or leg pain.The existence of one cause does not exclude the other.Priformis syndrome should not be a diagnosis of exclusion.

In the differential diagnosis of hip and/or leg pain, physical examination to exclude piriformis syndrome and injection of local anesthetic into the piriformis muscle is much less invasive than surgery to confirm lumbar spine pathology and can be performed as an outpatient.Thus, early diagnosis and appropriate treatment process is accelerated. If there is an unfavorable response to the local injection, investigation for lumbar vertebral pathologies can be initiated.

The purpose of the investigators under this information and justifications is; To determine the frequency of Priformis syndrome in patients presenting with hip and/or leg pain and to investigate the association of Priformis syndrome with other pathologies of the lumbar spine and hip.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with unilateral hip and/or leg pain

Exclusion Criteria:

* no

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
To determine the frequency of Priformis syndrome | 1 months
  Change in Pain Scores on Visual Analogue Scale scores at 24 hours before and after Priformis muscule injection